CLINICAL TRIAL: NCT05151302
Title: The Italian Version of the Computer-Vision Symptom Scale Questionnaire: Translation, Validation and Reliability.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Gemma Caterina Maria Rossi, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CVSS17
Record Dates: First submitted 2021-11-11; First posted 2021-12-09 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2022-03

CONDITIONS: Video Display Terminal Workers; Computer Vision Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- completion of the computer vision symptom scale questionnaire, italian version (Other): video display terminal (VDT) workers completed the questionnaire
  Interventions: Diagnostic Test: computer vision symptom scale (CVSS) questionnaire

INTERVENTIONS:
Diagnostic Test: computer vision symptom scale (CVSS) questionnaire — Subjects working at VDT for >20 hours a week and accessing to the Eye Clinic in order to complete an ocular examination and subjects working at the Foundation accessing to the Eye Clinic in order to complete an ocular status evaluation according to Italian Law 81/08 will be asked to self-complete the questionnaire in presence of the attending junior ophthalmologists prior to the visit with the Ophthalmologist, to avoid interference with visit results (communication of bad/good news)

SUMMARY:
Video display terminal users frequently refer computer-related visual and ocular symptoms, that are the most frequently occurring health problems among such these subjects.

The Italian law has established an eye examination to assess ocular status (D.Lgs 81/08 ex law 626/96) in VDT workers: subjects are evaluated by clinical signs and symptoms. The availability of a validated questionnaire could be very useful to diagnose visual disturbances and to follow them during follow-up examinations in 2014, a Spanish group has developed and validated a questionnaire for the assessment of visual and ocular symptoms in VDT workers.

Aim of the present study is to make available to Italian health professionals a new instrument to assess asthenopic symptoms, taking into account the patient's perspective.

ELIGIBILITY:
Inclusion Criteria:

* VDT workers as defined by the Italian law (>20 hours a week on PC); in the control group patients no VDT workers.
* VDT workers at the Foundation or VDT accessing to the general service of the Clinic for a routine visit (VDT group)
* patients, not working at VDT, accessing to the "general service" of the eye clinic to perform a routine visit will be asked to participate the study (control group)
* no ocular surgery in the preceding 6 months
* written consent to participate to study procedures and personal data utilization in an encoded form

Exclusion Criteria:

* ocular surgery in the preceding 6 months
* patients unable to respond to questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2015-02-11 (Actual); Primary Completion 2017-02-06 (Actual); Study Completion 2017-02-06 (Actual)

PRIMARY OUTCOMES:
To assess reliability (Cronbach alpha) of the CVSS | one year
  Cronbach alpha

SECONDARY OUTCOMES:
To assess: -item internal consistency -equality of item-scale correlations -item discriminant validity -temporal stability -discriminating ability (between VDT and non-VDT workers) -external validity | one year
  statistical examinations

CONTACTS AND LOCATIONS:
Overall Officials: Gemma Caterina M Rossi, Principal Investigator — irccs policlinico san matteo foundation

IPD SHARING:
Plan to Share IPD: No